CLINICAL TRIAL: NCT01980082
Title: Antibiotic Prophylaxis for Revision, Clean Head and Neck Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, yotam shkedy, Resident, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ProphylacticABxHN
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Surgical Wound Infection
Keywords: head and neck surgery; surgical wound infection; antibiotic prophylaxis
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefazolin (Active Comparator): Cefazolin
  1 gram/2 gram if body mass index > 40 - one time dose, 30-60 min prior to incision.
  Interventions: Drug: Cefazolin
- Placebo (Placebo Comparator): 1 dose of placebo - NaCl 0.9% with no drugs added to it.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cefazolin — Antibiotic
  Other Names: Cefamezine
  Arms: Cefazolin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
We hypothesized that revision clean head & neck surgery may have a higher rate of wound infection that may be lowered with prophylactic antibiotic treatment.

DETAILED DESCRIPTION:
Surgical wound infection (SWI) is a common complication in many operations, including head and neck (H&N) surgery, with reported rates ranging between 3.5 to 87%. While prophylactic antibiotic use has been shown to decrease SWI in clean-contaminated and contaminated surgery, its use in clean surgery is debatable. In most types of clean surgery the value of prophylactic antibiotics is minimal, however in some cases it might be justified, including in radical neck dissections, in a previously irradiated neck, those with a tracheostomy and immunosuppressed patients - although there is no consensus regarding these risk factors.

Previous research has shown that adherence to guidelines regarding prophylactic antibiotic use is lacking, with one study showing a greater than 40% rate of inappropriate antibiotic administration. This may be partially attributed to some patients having other risk factors, not covered by existing guidelines.

One such risk factor is previous H&N surgery. While there are no studies addressing this issue in H&N surgeries, a study in clean neurosurgical operations has shown an almost trice-fold increase in SWI rates in some operations (4% vs. 13%).

The purpose of this study is to investigate the effect of prophylactic antibiotic use in repeat clean H&N surgery.

This is a double-blind, randomized, placebo-controlled study. The study will be conducted at the Otolaryngology department in Rabin Medical Center, Petah Tikva.

Patients will be randomly assigned to 2 groups, with each group composed of 50 patients: a study group which will receive 1 dose of intravenous Cefazolin 1 gram/2 gram if body mass index > 40 or a control group which will receive 1 dose of placebo. The drug/placebo will be given 30-60 minutes prior to incision. Previous studies have shown no benefit for longer duration of prophylactic antibiotic coverage. Both the study drug and placebo will be prepared by a designated nurse from the department. The nurse will use a randomization site (www.random.org with min set to 1 and max set to 1000) to give each participant a number. A predefined Excel table will contain an assignment of each number to one of the groups. Only this nurse will know the assignment of each patient and she will not be assessing the patient post-operatively. The patients, surgeons and researchers will be blinded to the patients' assignments.

The status of the surgical wound will be assessed daily during hospitalization and again on the planned follow-up visit 3-4 weeks after discharge. During the follow-up visit, patients will be questions regarding symptoms and signs of SWI and antibiotic prescriptions given during the post-operative period.

SWI diagnosis will be according to the Center for Disease Control's "guideline for surgical site infection". Treatment of SWI will be according to regular department protocols (with no regard to study allocation).

ELIGIBILITY:
Inclusion Criteria:

* Previous H&N surgery.
* Planned second H&N clean surgery (the definition of a second H&N surgery is a surgery which will include the same skin incision as the previous operation).

Exclusion Criteria:

* Previous neck irradiation.
* Tracheostomy status.
* Immunosuppression.
* Concurrent infection which requires antibiotic use.
* Any other factor during the surgery which the surgeon estimates requires prophylactic antibiotic use.
* Allergy to cephalosporins and allergy to penicillin which precludes the use of cephalosporins (e.g. anaphylaxis).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-01; Primary Completion 2017-06-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Surgical wound infection, sepsis, bacteremia. | 1 month from surgery

SECONDARY OUTCOMES:
Length of stay | 1 month from surgery
  Length of post-operative stay
Drug-induced adverse reactions | 1 month from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yotam Shkedy, MD, Principal Investigator — Rabin Medical Center, Petach Tikva, Israel
Locations (1):
- Department of Otolaryngology, Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Simo R, French G. The use of prophylactic antibiotics in head and neck oncological surgery. Curr Opin Otolaryngol Head Neck Surg. 2006 Apr;14(2):55-61. doi: 10.1097/01.moo.0000193183.30687.d5. PMID 16552259
- [Background] Velanovich V. A meta-analysis of prophylactic antibiotics in head and neck surgery. Plast Reconstr Surg. 1991 Mar;87(3):429-34; discussion 435. PMID 1825518
- [Background] Seven H, Sayin I, Turgut S. Antibiotic prophylaxis in clean neck dissections. J Laryngol Otol. 2004 Mar;118(3):213-6. doi: 10.1258/002221504322927991. PMID 15068519
- [Background] Brown BM, Johnson JT, Wagner RL. Etiologic factors in head and neck wound infections. Laryngoscope. 1987 May;97(5):587-90. doi: 10.1288/00005537-198705000-00009. PMID 3573905
- [Background] Tenney JH, Vlahov D, Salcman M, Ducker TB. Wide variation in risk of wound infection following clean neurosurgery. Implications for perioperative antibiotic prophylaxis. J Neurosurg. 1985 Feb;62(2):243-7. doi: 10.3171/jns.1985.62.2.0243. PMID 3968563
- [Derived] Shkedy Y, Stern S, Nachalon Y, Levi D, Menasherov I, Reifen E, Shpitzer T. Antibiotic prophylaxis in clean head and neck surgery: A prospective randomised controlled trial. Clin Otolaryngol. 2018 Dec;43(6):1508-1512. doi: 10.1111/coa.13195. Epub 2018 Aug 14. PMID 30027615